CLINICAL TRIAL: NCT03318692
Title: Patient Specific Template Guided Pedicle Instrumentation Versus the Fluoroscopy Guided Free Hand Technique - a Randomized Prospective Trial
Brief Title: Patient Specific Template Guided Pedicle Instrumentation Versus Free Hand Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MySpine clinical
Record Dates: First submitted 2017-06-29; First posted 2017-10-24 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Spinal Fusion

STUDY DESIGN:
Intervention Model Description: prospective, randomized, partially blinded
Who Masked: Participant
Masking Description: Patient is masked to the surgery procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MySpine System (Experimental): pedicle screw implantation (spondylodesis) using the MySpine System. post surgery CT.
  Interventions: Procedure: spondylodesis; Procedure: CT
- free-hand (Active Comparator): Freehand (fluoroscopically controlled) implantation of pedicle screw (spondylodesis). Post surgery CT
  Interventions: Procedure: spondylodesis; Procedure: CT

INTERVENTIONS:
Procedure: spondylodesis — Dorsal instrumentation with transpedicular screws (spondylodesis)
Procedure: CT — CT of operated area is performed within 7 days of surgery

SUMMARY:
The clinically already tested and approved MySpine system is compared to the free-hand dorsal instrumentation, which is the gold standard in spondylodesis surgery. The aim of this study is to investigate whether or not the pedicle screw can be inserted anatomically more accurately by the MySpine system than by the conventional free-hand method using intraoperative fluoroscopy.

DETAILED DESCRIPTION:
Patients with an indication for spondylodesis are included according to the inclusion criteria and exclusion criteria. Subsequently, randomization into the MySpine and conventional group is performed. Patients remain blinded to the randomization.

On the basis of a computed tomography, the surgeon plans the entry points, the screw size and length, as well as the angle of the screws in two planes (sagittal and axial) on the computer. In the MySpine group, a three-dimensional, digital reconstruction of the spine is made using Medacta International SA software. On the basis of these planning files, three-dimensional templates with guide channels (guides) are produced for each individual vertebra. These guides can be applied dorsally to the bony anatomy and thus specify the entry points as well as the direction of the screw. Also, replicas of the individual vertebra are produced in the 3D printer.

The patients are operated in a prone position via a dorsal approach. After preparation of the dorsal process, vertebral arches and vertebral joints as well as the transverse process, the screws are implanted with one of the following methods depending on the randomization:

1. Freehand (fluoroscopically controlled)
2. MySpine System

Postoperatively, all patients undergo computed tomography of the operated area. On the basis of this computed tomography the number of pedicle perforations as well as their extent should be determined according to the simplified Laine classification. These results are to be statistically evaluated with the question of whether there are significant differences between the two techniques with respect to the absolute and individual number of pedicle perforations, as well as their extent. It is also to be examined whether these results show a dependence on the level of experience of the surgeon.

In addition to the individual radiation exposure (cumulative irradiation time in seconds and irradiation dose in cGy), the time for the dorsal instrumentation for each of the two systems per surgeon is also to be measured and evaluated.

In the follow-up, the outcome is also recorded by means of pain registration, ODI score and complication detection (infections, pedicle fractures, implant loosening, pseudoarthrosis, re-operations).

The follow-up assessments 6 weeks, 6 months, 1 year and 2 years after surgrey are peformed according to institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* Indication for spondylodesis independent of the study
* Signed consent
* Male and female patients aged 18 years and over

Exclusion Criteria:

* Polyamide-PA 12 allergy
* Pregnant or lactating women
* Known or suspected non-compliance with the protocol, drug or alcohol abuse
* inability of the patient to follow the trial procedure, e.g. Due to language problems, mental illness, dementia
* Prior participation in the clinical Trial
* Inclusion of the test person, his / her family members, employees or other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
accuracy | within 7 days post surgery
  Anatomical accuracy of pedicle screw implantation (intactness of the pediculate cortex in 3 planes), postoperatively measured via computertomographically existing or nonexisting pedicle perforation and their extent according to the simplified Laine classification: Grade A (<2 mm), Grade B (2-4 mm) and Grade C (> 4 mm)

SECONDARY OUTCOMES:
duration | during surgery
  Intraoperative time spent on dorsal Instrumentation is documented and compared between the groups
Radiation exposure | during surgery
  cummulative Radiation exposure during surgery is measured and compared between the groups
blood loss | during surgery
  blood loss during surgery is documented and compared between the groups
complications | during surgery until end of follow up (24 months after surgery)
  intraoperative and post-operative complications such as pedicle fractures, implant loosening, infections and pseudo arthrosis are documented and compared between the groups
reoperations | until end of follow up (24 months after surgery)
  reoperations are documented and compared between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Farshad, Prof. Dr.med., Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
IPD only available to study personnel. statistical Analysis will be done with encoded data only. study results will be published